CLINICAL TRIAL: NCT05343273
Title: Total, Free, and Bioavailable 25-Hydroxyvitamin D Levels in Patients With Periodontitis (Stage III): A Case-Control Study
Brief Title: 25-Hydroxyvitamin D Levels in Patients With Periodontitis (Stage III)
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Tugba Aydin, Assistant Professor, Ataturk University
Other Study IDs: 9099
Record Dates: First submitted 2022-04-07; First posted 2022-04-25 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Vitamin D Deficiency; Periodontitis
Keywords: Total 25(OH)D; Bioavailable 25(OH)D; Free 25(OH)D; Periodontitis
MeSH Terms: conditions — Vitamin D Deficiency; Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

GROUPS / COHORTS (2):
- Healthy
  Interventions: Diagnostic Test: taking a blood sample
- Periodontitis
  Interventions: Diagnostic Test: taking a blood sample

INTERVENTIONS:
Diagnostic Test: taking a blood sample — blood collection for routine biochemical analysis

SUMMARY:
Periodontitis; is an inflammatory disease of tissues characterized by bone destruction around the teeth. Vitamin D plays an important role in several inflammatory diseases by promoting the expression of inflammatory cytokines such as interleukin IL-1, IL-6, and IL-1β, which are directly related to periodontal attachment loss and bone demineralization. These facts suggest that vitamin D may be associated with periodontal disease. Many studies have been conducted on the relationships between serum 25-hydroxyvitamin D (25(OH)D) levels, periodontal disease, and tooth loss. However, as far as we know, there is no study on the relationship between periodontitis and free and bioavailable 25 (OH) vitamin D. In our study, over the age of 35; two groups will be formed, consisting of 40 healthy and 40 periodontitis individuals. Serum total 25 (OH) D level and vitamin D binding protein level will be analyzed by ELISA method, and bioavailable 25 (OH) D level will be calculated using total 25 (OH) D and vitamin D binding protein levels. The aim of this study; To evaluate the total, free and bioavailable 25 (OH) vitamin D levels of patients with periodontitis by comparing them with healthy controls, and to investigate whether bioavailable 25 (OH) D plays a role in the pathogenesis of periodontitis or can be a simple marker of disease activity in the light of these findings.

ELIGIBILITY:
Inclusion Criteria:

* Without systemic disease,
* Had a least 14 teeth

Exclusion Criteria:

* Individuals with a history of systemic or topical oral antimicrobial therapy use in the last 3 months,
* Individuals with an allergy to any ingredient used in the study,
* Smokers,
* Pregnant or breastfeeding women,
* Using vitamin D,
* Individuals diagnosed with obesity

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Forty patients with stage 3 periodontitis and 40 healthy volunteers were included in this case-control study at Atatürk University, Department of Dentistry, Department of Periodontology.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Measurements of 25(OH)D | Within one week of collecting blood samples from all participants.
  Total 25(OH)D levels in serum samples will be measured by ELISA method, using the "Human 25-Dihydroxy vitamin D ELISA Kit" (BT LAB, Cat No: E1981Hu, China) in accordance with the manufacturer's instructions. Results will be recorded in ng/mL.
Measurements of VDBP | Within one week of collecting blood samples from all participants.
  VDBP levels in serum samples will be studied by ELISA (Enzyme Linked Immunosorbend Assay) method using Elabscience brand kit (Elabscience Biotechnology Co., Ltd). Results will be recorded in (ug/mL.
Measurements of Albumin | Within one week of collecting blood samples from all participants.
  Serum albumin levels (g/dL) will be measured on the Roche Cobas c702 instrument (Germany) using commercial kits.
Calculation of Bioavailable 25(OH)D | Within one week of collecting blood samples from all participants.
  It will be calculated using calculations using affinity constants and calculated free 25(OH)D and measured albumin levels.
  Kalb = affinity constant between vitamin D and albumin = 6 x 10^5 M^-1
  Bioavailable 25(OH)D concentration = (6 x 10^5 x [Albumin]+1) x calculated free 25(OH)D
  Results will be recorded in ng/mL.
Calculation of Bioavailable Free 25(OH)D | Within one week of collecting blood samples from all participants.
  It will be calculated using calculations using affinity constants and measured total serum 25(OH)D, VDBP and albumin levels.
  Kalb = affinity constant between vitamin D and albumin = 6 x 10^5 M^-1 KVDBP = affinity constant between vitamin D and VDBP = 7 x 10^8 M^-1 [Albumin] = serum albumin concentration = (serum albumin g/L) / 66.430 g/mol [VDBP] = serum vitamin D binding protein concentration = (serum VDBP g/L) / 58.000 g/mol
  Free 25(OH)D concentration = Total 25(OH)D / 1+(6 x 10^5 x [Albumin]) + (7 x 10^8 x [VDBP])
  Results will be recorded in pg/mL.

SECONDARY OUTCOMES:
Dental Plaque | Day 1
  Plaque scores recorded by using the Silness&Löe Plaque Index
  PI 0: No observable plaque PI 1: A thin film of plaque is detected at the gingival margin by running a probe or explorer across the tooth surfaces PI 2: A moderate amount of plaque is detected along the gingival margin. Plaque is visible clinically.
  PI 3: Heavy plaque accumulation is detected at the gin- gival margin and in the interdental spaces.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, None Selected, Turkey (Türkiye)

REFERENCES:
- [Derived] Aydin T, Dilsiz A, Eminoglu DO, Sahin AB, Laloglu E, Bayrakdar YE. Total, free, and bioavailable 25-hydroxyvitamin D levels in patients with periodontitis (stage III): a case-control study. Clin Oral Investig. 2023 Jan;27(1):421-430. doi: 10.1007/s00784-022-04844-9. Epub 2023 Jan 4. PMID 36598602